CLINICAL TRIAL: NCT03983655
Title: Effect of High Frequency/Low Intensity Transcranial Magnetic Stimulation in Cognitive Traits of an Elderly Population of Subjects With Mild Cognitive Impairment and Mild Dementia: A Randomized, Double Blind, Parallel Group, Sham Controlled Clinical Trial
Brief Title: Effect of High Frequency/Low Intensity Transcranial Magnetic Stimulation in Cognitive Traits of an Elderly Population of Subjects With Mild Cognitive Impairment and Mild Dementia.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Actipulse Neuroscience (Unknown)
Responsible Party: Principal Investigator, Alberto José Mimenza Alvarado, Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: GER-2962-19-20-1
Record Dates: First submitted 2019-05-21; First posted 2019-06-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Mild Cognitive Impairment; Mild Dementia
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real High Frequency Low Intensity TMS (Experimental): Two sessions of transcranial magnetic stimulation each day for 6 monts. The coil of the device emits a pulsed magnetic field at an aproximate frequency of 125 hz and an intensity of 10 gauss.
  Interventions: Device: High Frequency Low Intensity TMS
- Sham High Frequency Low Intensity TMS (Sham Comparator): Two sessions of transcranial magnetic stimulation each day for 6 monts. The coil of the device does not emit a magnetic field.
  Interventions: Device: High Frequency Low Intensity TMS

INTERVENTIONS:
Device: High Frequency Low Intensity TMS — 125 hz, 10 gauss, 2 times daily for 6 monts

SUMMARY:
There are no pharmacological interventions that delay or prevent the transition of mild cognitive impairment to dementia. Several studies have shown that transcranial magnetic stimulation (TMS) could be useful in increasing cognitive traits in dementia.

As TMS is performed in a clinical setting, transportation, mobility and high costs of treatment, limit the number of TMS sessions dementia patients can receive. Most of the trials do not apply more than 20 TMS sessions

Here, a randomized, sham controlled, paralallel group, clinical trial will be performed in order to asess the efficacy at improving cognitive traits of a novel TMS device that uses high frequency and low intensity pulses. As the device is portable and can be used from home without clinical supervision, the stimulation will be applied two times per day for a period of 6 months.

ELIGIBILITY:
IInclusion Criteria:

( - ) CDR less or equal to 1 ( - ) Mild cognitive impairment by Petersen criteria ( - ) Conserved or corrected sight ( - ) Enrolled at INCMNSZ for medical care ( - ) Be able to read and write ( - ) Willing and able to provide written informed consent

Exclusion Criteria:

( - ) Other neurodegenerative disorder different than mild cognitive impairment or mild dementia ( - ) Metabolic disease without medical care ( - ) Epilepsy ( - ) Deep brain stimulator ( - ) Metalic prosthethics in the skulls ( - ) Major depressive disorder ( - ) Previous utilization of other neuromodulation technique ( - ) Signs or symptoms of increased intracraneal pressure

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2020-05-17 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients suffering any kind of adverse effect | 6 months

SECONDARY OUTCOMES:
Change from baseline of total Katz Index of Independence in Activities of Daily Living at 3 months | 3 months
Change from baseline of total Katz Index of Independence in Activities of Daily Living at 6 months | 6 months
Change from baseline of total Lawton Instrumental Activities of Daily Living Scale at 3 months | 3 months
Change from baseline of total Lawton Instrumental Activities of Daily Living Scale at 6 months | 6 months
Change from baseline of total Geriatric Depression Scale at 3 months | 3 months
Change from baseline of total Geriatric Depression Scale at 6 months | 6 months
Change from baseline of total Montreal Cognitive Assessment at 3 months | 3 months
Change from baseline of total Montreal Cognitive Assessment at 6 monts | 6 months
Change from baseline of total Frontal Asessment Battery at 3 monts | 3 months
Change from baseline Frontal Asessment Battery at 6 monts | 6 months
Change from baseline ADAS-COG at 6 monts | 6 months
  Alzheimer´s Disease Assessment Scale-Cognitive

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mimenza-Alvarado AJ, Aguilar-Navarro SG, Martinez-Carrillo FM, Rios-Ponce AE, Villafuerte G. Use of Fast Gamma Magnetic Stimulation Over the Left Prefrontal Dorsolateral Cortex for the Treatment of MCI and Mild Alzheimer's Disease: A Double-Blind, Randomized, Sham-Controlled, Pilot Study. Front Neurol. 2021 Sep 9;12:729872. doi: 10.3389/fneur.2021.729872. eCollection 2021. PMID 34566873